CLINICAL TRIAL: NCT05506293
Title: European Multicentre Registry of Percutaneous Paravalvular Leak Closure - EuroPVL Study
Brief Title: European Multicentre Registry of Percutaneous Paravalvular Leak Closure
Acronym: EuroPVL
Status: Recruiting | Type: Observational
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Collaborators: Easy-CRF (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019-A02930-57
Record Dates: First submitted 2022-03-07; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Cardiac Valve Disease; Paravalvular Aortic Regurgitation; Paravalvular Mitral Regurgitation; Paravalvular Leak; Quality of Life; Outcomes
Keywords: paravalvular leak; percutaneous intervention; quality of life; outcomes
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- paravalvular leak: patients referred for percutaneous paravalvular leak closure
  Interventions: Procedure: percutaneous paravalvular leak closure

INTERVENTIONS:
Procedure: percutaneous paravalvular leak closure — the procedure consists of deployment of an occluder or a vascular plug within the cardiac paravalvular leak. The device is inserted percutaneously from a femoral vascular approach or from a trans-apical approach. The device is deployed through a delivery sheath within the leak. Stability and efficacy to occlude the leak are assessed by transoesophageal echocardiography prior to device release.
  Type of devices to be inserted varied :
  * Amplatzer vascular plug 3
  * occlutech paravalvular leak device
  * amplatzer vascular plug 2
  * amplatzer muscular ventricular septal defect
  * amplatzer vascular plug 4
  Devices to be implanted are under the responsability of the local investigator and are not based on the study design.
  Other Names: transcatheter paravalvular leak closure

SUMMARY:
Paraprosthetic cardiac valve leaks are a progressive complication after after surgical or percutaneous heart valve replacement. These leaks can lead to heart failure and/or life-threatening hemolysis.

Percutaneous closure of para-prosthetic leaks has been developed as an alternative to surgery in high-risk patients. These procedures remain technically challenging with a significant risk of failure and complications, but this risk is improved since the development of dedicated prostheses and the increased experience of the operators. The data in the literature concerning percutaneous leak closure remain limited and disparate and mostly retrospective.The impact of the procedures on the quality of life of patients is not known. Beyond the technical aspects and the follow-up of major cardiovascular events, investigators also wonder what is the impact of these procedures on the quality of life of patients. Investigators hypothesize that even a partial reduction in paraprosthetic leakage may be associated with an improvement in quality of life through reduction of transfusion needs and/or reduction of dyspnea. A prospective study is warranted to assess the technical and clinical and clinical results of these procedures, together with the evaluation of the the possible benefit on the quality of life of the patients.

DETAILED DESCRIPTION:
OBJECTIVES OF THE STUDY MAIN OBJECTIVE To evaluate the clinical results of the transcatheter closure of para-prosthetic leaks.

SECONDARY OBJECTIVE Technical success of the procedure defined by successful placement of the prosthesis at the intended site with at least a 1 grade reduction in leakage and residual leakage grade 0-1 Change in quality of life after closure of para-prosthetic leakage at 3 months Evolution of clinical and biological markers of hemolysis and heart failure between at 3 months evolution of clinical markers of functional capacity 4. JUDGMENT CRITERIA 4.1 PRIMARY ENDPOINT

-Clinical success of the procedure:

Clinical success will be assessed on a composite endpoint at 2 years:

* vital status,
* hospitalization for heart failure,
* blood transfusion for hemolysis,
* surgical or percutaneous re-intervention on the treated valve. 4.2 SECONDARY ENDPOINTS The technical, echographic, biological and clinical data of the procedure and post procedure will be recorded as well as the complication rates. The EQ5D-5L quality of life score will be evaluated before the procedure, between 1 and 3 months, and post procedure.

STUDY POPULATION INCLUSION CRITERIA

To be included, each patient must meet all of the following conditions:

* Patients aged 16 years and older,
* Patients or the representative of the parental authority of the minor patient who does not object to participation in the observatory,
* Patients referred for a para-prosthetic leak closure procedure NON-INCLUSION CRITERIA Patients presenting at least one of the following criteria cannot be included
* Patients under 16 years of age,
* Refusal of the patient or the representative of the parental authority of the minor patient to participate in the observatory.

ELIGIBILITY:
Inclusion Criteria:

* ≥16 years of age No opposition from the patient or the representative of the parental authority if the patient is a minor Patient referred for a percutaneous paraprosthetic leak closure procedure

Exclusion Criteria:

* < 16 years old Refusal of the patient to participate in the observatory or of the legal representative if the patient is a minor

Ages: 16 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Included patients are included as part of their routine clinical care. The percutaneous intervention is not indicated for the purpose of the study but according to each centre policy after a medico-surgical meeting.
  Prior to percutaneous intervention, a large investigation of functional status, quality of life, biological exam and echocardiography is performed. This investigation is done again at 1 and 2 years
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
clinical success | 1 year
  Device success is a composite criteria including all of the following conditions:
  No rehospitalizations or reinterventions for hemolysis No rehospitalizations or reinterventions for Heart Failure Improvement versus baseline in symptoms defined as decrease in NYHA functional class of at least one class vs. baseline

SECONDARY OUTCOMES:
clinical success | 2 year
  Clinical success will be assessed on a composite endpoint at 2 years including the following conditions:
  * no death
  * no hospitalization for heart failure,
  * no blood transfusion for hemolysis,
  * no surgical or percutaneous re-intervention on the treated valve.
quality of life | 30 days
  evolution of quality of life between baseline and 3 months after the procedure on the EQ5D-5L score

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Hascoet, MD, PhD, Principal Investigator — s.hascoet@ghpsj.fr
Locations (33):
- CHU Charleroi, Charleroi, Belgium
- Podlesi hospital, Třinec, Czechia
- France (21):
  - CHU Amiens, Amiens
  - Hopital d Annecy, Annecy
  - CHU Henri Mondor, Créteil
  - CHU Grenoble, Grenoble
  - centre chirurgical Marie Lannelongue, Le Plessis-Robinson
  - Hopital Prive Brabois, Lille
  - CHU La Timone, Marseille
  - Hopital Europeen, Marseille
  - Hopital Prive Clairval, Marseille
  - CHU Nancy, Nancy
  - Hopital prive les Franciscaines, Nîmes
  - HEGP, Paris
  - Hopital Bichat, Paris
  - Hopital Pitie Salpetriere, Paris
  - CHU Rennes, Rennes
  - Hopital Charles Nicolle, Rouen
  - Centre Cardiologique du Nord, Saint-Denis
  - institut Arnault Tzanck, Saint-Laurent-du-Var
  - CHU Toulouse, Toulouse
  - Clinique Pasteur, Toulouse
  - Medipole Lyon Villeurbanne, Villeurbanne
- National and kapodistrian university of athens, Athens, Greece
- University School of Milan, Milan, Italy
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Vilnius University Hospital, Vilnius, Lithuania
- hospital infantil de Mexico Frederico Gomez, Mexico City, Mexico
- Medical University of Silesia, Katowice, Poland
- Hospital Clinic of Barcelona, Barcelona, Spain
- Kocaeli University Medical Faculty, Kocaeli, Turkey (Türkiye)
- United Kingdom (2):
  - Royal Papworth hospital, Cambridge
  - Edinburgh Royal Infirmary, Edinburgh

IPD SHARING:
Plan to Share IPD: No